CLINICAL TRIAL: NCT05649891
Title: Clinical Use of an Emergency Manual by Resuscitation Teams and Impact on Performance in the Emergency Department
Brief Title: Checklists Resuscitation Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01896-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Shortness of Breath; Chest Pain; Abdominal Pain; Altered Mental Status; Syncope; Seizures; Vertigo; Trauma; Allergic Reaction; Fever; Cardiac Arrest; Asthma Acute; COPD Exacerbation Acute; Pneumonia; Pulmonary Edema - Acute; Bradycardia; Tachycardia; Shock; Burns; Poisoning; Diabetic Ketoacidosis; Hyperglycemic Hyperosmolar Nonketotic Syndrome
MeSH Terms: conditions — Dyspnea; Chest Pain; Abdominal Pain; Syncope; Seizures; Vertigo; Wounds and Injuries; Hypersensitivity; Fever; Heart Arrest; Pneumonia; Bradycardia; Tachycardia; Shock; Burns; Poisoning; Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients managed with Emergency Manual access (Experimental): Consecutive priority 1 patients managed by resuscitation teams with access to an Emergency Manual
  Interventions: Other: Emergency Manual

INTERVENTIONS:
Other: Emergency Manual — Collection of crisis checklists and fact sheets

SUMMARY:
The study will systematically evaluate how an emergency manual-a collection of checklists and fact sheets-affects the performance of resuscitation teams during the management of priority one patients in an emergency department.

DETAILED DESCRIPTION:
Simulation-based studies indicate that crisis checklist use improves management of patients with critical conditions in the emergency department (ED). This six-month-long study prospectively evaluates a digital emergency manual-a collection of crisis checklists and fact sheets-during the management of priority 1 patients in the Skåne University Hospital at Lund's ED.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive priority 1 patients managed in the resuscitation room of Skåne University Hospital at Lund's Emergency Department

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Degree of indication of interventions performed thanks to Do-Confirm Emergency Manual use | 1 hour
  The primary outcome measures are the proportions of interventions performed thanks to Do-Confirm EM use graded as indicated, of neutral relevance, and not indicated.

SECONDARY OUTCOMES:
Team's subjective evaluation of Emergency Manual value | 1 hour
  The team's subjective evaluation of the EM's value is recorded prior to the logging out from the EM using a Likert scale of 1 to 6.
Degree of indication of interventions that might have been performed had the Emergency Manual been used | 1 hour
  Fifty patients that presented during the six-month period preceding EM implementation, are identified. These 50 patients are selected based on matching to the 50 patients where the EM was used, using age, presenting complaint and relevant co-morbidities. In addition, fifty patients where the EM was not used during the pilot study period are also identified based on the same matching process. The EM is accessed to determine whether additional interventions would have been performed, had the EM been used. All interventions-those actually performed as well as those that might have been performed had the EM been used-are then assessed for degree of indication by three external reviewers.
Structured interviews | Up to 8 weeks
  Teams can electronically request contact with the investigators to report specific events related to EM use. If so, the following data is extracted during a structured interview:
  * patient age, sex, presenting complaint and suspected diagnosis
  * seniority of the physician initially in charge of the case
  * events or concerns relating to EM use
  * mode of EM use (Do-Confirm, Read-Do, Sampling) and sections relevant to the case
  * personnel's assessment of the impact of the EM on patient care
  * personnel's assessment of impact of the EM on team members and teamwork
  * personnel's suggestions for EM improvement

CONTACTS AND LOCATIONS:
Overall Officials: Eric Dryver, MD, Principal Investigator — Skane's University Hospital in Lund, Emergency Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dryver E, Olsson de Capretz P, Mohammad M, Armelin M, Dupont WD, Bergenfelz A, Ekelund U. Clinical use of an emergency manual by resuscitation teams and impact on performance in the emergency department: a prospective mixed-methods study protocol. BMJ Open. 2023 Oct 17;13(10):e071545. doi: 10.1136/bmjopen-2022-071545. PMID 37848292